CLINICAL TRIAL: NCT00638222
Title: Carvedilol and Micro T-Wave Alternans in Hypertensives With Chronic Kidney Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Christopher Cooper, MD, Professor, Interim Chair/Dir Cardiovas Research Cntr, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UTHSC-08
Record Dates: First submitted 2008-03-05; First posted 2008-03-19 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Vascular Disease; Kidney Disease
Keywords: Carvedilol; Heart Disease; Vascular Disease; Kidney
MeSH Terms: conditions — Vascular Diseases; Kidney Diseases; Heart Diseases | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Study Participants (Active Comparator): All enrolled participants were randomized to receive Carvedilol or Placebo in a 2-way crossover design. Each intervention was administered over 8 weeks before switching to the alternative intervention. The study was terminated early, and data were not unblinded so participants cannot be reported separately.
  Interventions: Other: Carvedilol and Placebo

INTERVENTIONS:
Other: Carvedilol and Placebo — All enrolled participants were randomized to receive Carvedilol or Placebo in a 2-way crossover design. Each intervention was administered over 8 weeks before switching to the alternative intervention. The study was terminated early, and data were not unblinded so participants cannot be reported separately.

SUMMARY:
Evaluate effectiveness of Carvedilol CR on Micro T-Wave Alternans in high risk hypertensives

DETAILED DESCRIPTION:
The effect of Carvedilol CR on Micro T-Wave Alternans will be assessed in 30 hypertensives with stage 4 or 5 chronic kidney disease utilizing a cross-over design and contrasting no treatment against active treatment periods of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older
* Chronic kidney disease
* Must be able to do stress test

Exclusion Criteria:

* Must not be mentally disabled
* Unable to provide informed consent
* Unable or unwilling to comply with study protocol or procedures
* Pregnancy or unknown pregnancy status in female of childbearing potential
* Participation in any drug trial during the study period
* Prior enrollment in this study
* Active liver disease
* Currently on β-blocker medication at the time of enrollment
* Known history of asthma exacerbation with β-blocker therapy
* Second or third degree AV nodal block or bradycardia with resting heart rate <50 bpm
* Prior allograft organ transplantation
* Planned allograft transplantation reasonably foreseen within the active treatment period
* Electrocardiographic left or right bundle branch block
* Permanent implanted pacemaker
* Atrial fibrillation
* Ongoing treatment with any of the following medications: sotalol (Betapace), azimilide (Stedicor), quinidine (Quinidex), disopyramide (Norpace), dofetilide (Tikosyn), ibutilide (Corvert), procainamide (Procanbid), bepridil (Vascor), amiodarone (Cordarone), clarithromycin (Biaxin), erythromycin (Eryc), halofantrine (Halfan), pentamidine (Pentam), sparfloxacin (Zagam), domperidone (Motilium), droperidol (Inapsine), chlorpromazine (Thorazine), haloperidol (Haldol), mesoridazine (Serentil), thioridazine (Mellaril), pimozide (Orap), arsenic trioxide (Trisenox), cisapride (Propulsid), lidoflazine (Clinium), and methadone (Dolophine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cooper,, MD, Principal Investigator — University of Toledo
Locations (2):
- United States (2):
  - University of Toledo, Health Science Campus, Toledo, Ohio
  - Site Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Carvedilol Then Placebo: Subject will receive Carvedilol over 8 weeks then receive Placebo for the 8 weeks following.
  Carvedilol: Subject will receive Carvedilol over 8 weeks then receive Placebo for the 8 weeks following.
- Placebo Then Study Drug: Subjects will receive placebo for 8 weeks then be given study drug for 8 more.
  Placebo: Subjects will receive placebo for 8 weeks then be given study drug for 8 more.
- All Participants: All enrolled participants were randomized to receive Carvedilol or Placebo in a 2-way crossover design. Each intervention was administered over 8 weeks before switching to the alternative intervention. The study was terminated early, and data were not unblinded so participants cannot be reported separately
Period: Overall Study
Arm/Group | Carvedilol Then Placebo | Placebo Then Study Drug | All Participants
Started | 0 | 0 | 6
Completed | 0 | 0 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carvedilol Then Placebo | Placebo Then Study Drug | All Study Participants | Total
Number analyzed (Participants) | 0 | 0 | 6 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] |  |  | 55 (15) | 55 (15)
Age, Categorical [Number; unit: participants]
  <=18 years |  |  | 0 | 0
  Between 18 and 65 years |  |  | 4 | 4
  >=65 years |  |  | 2 | 2
Gender [Number; unit: participants]
  Female |  |  | 0 | 0
  Male |  |  | 6 | 6
Region of Enrollment [Number; unit: participants]
  United States |  |  | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Micro T- Wave Alternans
Time Frame: week 1, 8, 11, 18
Arm/Group | Carvedilol Then Placebo | Placebo Then Study Drug
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Oxidized LDL
Time Frame: week 1, 8, 11, 18
Reporting Status: Not Posted

3. Secondary Outcome: Interleukin-6
Time Frame: week 1, 8, 11, 18
Reporting Status: Not Posted

4. Secondary Outcome: Plasma C-reactive Protein
Time Frame: week 1, 8, 11, 18
Reporting Status: Not Posted

5. Secondary Outcome: Plasma Cardiac Troponin T
Time Frame: week 1, 8, 11, 18
Reporting Status: Not Posted

6. Secondary Outcome: Plasma NT-pro BNP
Time Frame: week 1, 8, 11, 18
Reporting Status: Not Posted

7. Secondary Outcome: Plasma F2-isoprostanes
Time Frame: week 1, 8, 11, 18
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Carvedilol Then Placebo | Placebo Then Study Drug | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 2/6
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol Then Placebo (N=0) | Placebo Then Study Drug (N=0) | All Study Participants (N=6)
Low Blood Pressure (Cardiac disorders) | 0 | 0 | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carvedilol Then Placebo (N=0) | Placebo Then Study Drug (N=0) | All Study Participants (N=6)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Fluid Retention (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Shortness of Breath (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
Headache (General disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Cough (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain at Dialysis Catheter Site (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Right Groin Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Lower Extremity Angiogram (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dialysis Catheter Placed (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to poor enrollment leading to small number of subjects to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes